CLINICAL TRIAL: NCT00452179
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Cross-Over Study to Evaluate the Effects of APD125 in Patients With Chronic Primary Insomnia
Brief Title: Safety and Efficacy Study of APD125 in Patient With Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APD125-004
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Insomnia
Keywords: Sleep maintenance; Insomnia; Sleep Consolidation; Sleep; Insomnia, primarily sleep maintenance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Drug: APD125

SUMMARY:
The purpose of this study is to determine the effects of APD125 in patients with sleep maintenance insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Primary insomnia as defined in DSM-IV-TR, with predominant complaint of impaired sleep maintenance and confirmed by PSG
* PSQI >/= to 5
* Qualifying screening PSG parameters
* Generally good health

Exclusion Criteria:

* History of any sleep disorder, other than primary insomnia (e.g., restless leg syndrome, narcolepsy, sleep apnea, and disorders of REM/NREM sleep)
* Any clinically significant medical condition, laboratory finding, or ECG finding
* Pregnant and/or lactating females
* History of substance abuse within 2 years or positive urine drug screen
* Positive Hepatitis B/C results or HIV markers
* Apnea-Hypopnea Index (AHI) or a Periodic Limb Movement Arousal Index (PLMAI) > 10 as determined by screening PSG
* History of treatment with an investigational drug within the last month
* Recent travel involving crossing more than 3 time zones or plans to travel to another time zone (> 3 time zones) during the study

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Conventional PSG parameters

SECONDARY OUTCOMES:
Patient reported subjective sleep parameters

CONTACTS AND LOCATIONS:
Overall Officials: Warren A Prosser, Study Director — Arena Pharmaceuticals
Locations (1):
- San Diego, California, United States

REFERENCES:
- See also: Arena Pharmaceuticals Home Page — http://www.arenapharm.com